CLINICAL TRIAL: NCT00134368
Title: Pilot, Investigator-Initiated, Proof-of-Concept, Study of the Efficacy and Safety of Etanercept (Enbrel) in Adults With Vitiligo
Brief Title: Study of the Efficacy and Safety of Etanercept in Adults With Vitiligo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4489
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2008-08-07 (Estimated); Status verified 2008-08

CONDITIONS: Vitiligo
Keywords: vitiligo; etanercept
MeSH Terms: conditions — Vitiligo | interventions — Etanercept

INTERVENTIONS:
Drug: Etanercept

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of etanercept in adults with vitiligo.

DETAILED DESCRIPTION:
Subjects will self-administer etanercept 50 mg SQ twice weekly for 6 months. Lesion repigmentation will be evaluated at monthly visits.

ELIGIBILITY:
Inclusion Criteria:

* Vitiligo patients aged 18 years and older
* Vitiligo patients with evaluable lesions; duration of 3 months to 10 years.
* Disease interferes significantly with quality of life and/or involving 3% or more body surface area
* Subjects must have a negative tuberculin (TB) skin test at entry into the study
* If subject is a female of childbearing potential, she must agree to use adequate contraception (adequate contraception can include abstinence) and must have a negative serum pregnancy test the day of administration of study medication.
* If subject is a male and has reached puberty, he must agree to use adequate contraception during the study and for 1 month after discontinuation from study.
* Subject or designee must have the ability to self-inject investigational product or have a care giver at home who can administer subcutaneous injections
* Subject must be able to give informed consent; must authorize release and use of protected health information; and, if applicable, must assent to participate prior to enrollment to this study.

Exclusion Criteria:

* Unable to consent
* History of non-compliance with other therapies
* Concurrent therapy for vitiligo
* Systemic or photo-therapy within 4 weeks
* Topical therapy within 2 weeks
* Any medical condition in which etanercept would be contraindicated
* Any internal malignancy within 5 years (fully excised cutaneous, basal cell carcinoma or squamous cell carcinoma are exceptions)
* Pregnancy, not practicing effective birth control, or inability to practice safe sex during the length of the study.
* Lactation
* History of alcohol or drug abuse one year before and during the study.
* Any participation in another investigational drug study during the 4 weeks preceding this study.
* Known HIV-positive status; known history of any other mycobacterial disease or any other immuno-suppressing disease.
* Presence of a grade 3 or 4 infection < 30 days prior to the screening visit; between the screening visit and the first day of treatment on study; or any time during the study that, in the opinion of the Investigator, would preclude participation in the study.
* Patients should not receive live vaccines for 3 months prior to, or while on, study.
* A prior history of tuberculosis, and/or a positive PPD skin test and positive CXR at screening.
* Patients with previous or current exposure to any of the following TNF antagonists:

  * etanercept (Enbrel);
  * adalimumab (Humira); or
  * infliximab (Remicade).

These patients will not be eligible, even with a wash-out. Patients with previous or current exposure to Kineret will NOT be eligible, even with a wash-out. However, patients with prior or current exposure to biologics directed against T-cells (e.g. alefacept, efalizumab, siplizumab, etc.) will be eligible for enrollment into the study after a wash-out period of 4 weeks before first dose of study drug (baseline visit). It has to be protocol specific also.

* The subject has, in the Investigator's opinion, a chronic, severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, pulmonary, cardiovascular (congestive heart failure [CHF] of any severity; myocardial infarction [MI], cerebrovascular accident [CVA] or transient ischemic attack [TIA] within 3 months of screening visit; unstable angina pectoris; uncontrolled hypertension [sitting systolic blood pressure (BP) < 80 mm Hg or > 160 or diastolic BP > 100 mm Hg]), or neurological disease; known systemic lupus erythematosus (SLE); diabetes; or any other concomitant medical condition that places the participant at risk by participating this study and/or that may interfere with the conduct of the study.
* Chronic hepatitis B or hepatitis C, SLE, history of multiple sclerosis, transverse myelitis, optic neuritis or epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-11; Study Completion 2007-12

PRIMARY OUTCOMES:
Percent of subjects achieving 50% or more repigmentation at 6 months (Good or better on Physician's Global Assessment [PGA] score)

SECONDARY OUTCOMES:
Percentage of subjects achieving 75% or more repigmentation at 6 months (Excellent or better on PGA score)
Patient-Generated Global Assessment
Skin texture assessment

CONTACTS AND LOCATIONS:
Overall Officials: Alice Gottlieb, MD, PhD, Principal Investigator — UMDNJ-RWJMS
Locations (1):
- UMDNJ Psoriasis Center of Excellence, New Brunswick, New Jersey, United States